CLINICAL TRIAL: NCT03096379
Title: Differentiating Gut Tuberculosis and Crohn's Disease Via Magnetic Resonance Enterography
Brief Title: MRI Differentiating Gut TB and Crohn's
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Wai-Kay Seto, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: MRE-TB-CD
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Crohn Disease; Intestinal Tuberculosis
Keywords: TB; CD; MRE; ileocecal
MeSH Terms: conditions — Crohn Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Magnetic resonance imaging: Patients with new-onset of lower gastrointestinal symptoms and ileocecal mucosal lesions of uncertain diagnosis as evidenced by the presence of inflammation, ulceration, strictures or nodules on colonoscopy.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Enterography performed via magnetic resonance imaging

SUMMARY:
It is clinically challenging to differentiate Crohn's disease from gut tuberculosis especially in regions endemic of tuberculosis infection. The investigators plan to perform magnetic resonance enterography (MRE) who presented to our hospital in Shenzhen, China for new onset of lower gastrointestinal symptoms and ileocecal mucosal lesions of uncertain diagnosis as evidenced by the presence of inflammation, ulceration, strictures or nodules on colonoscopy. MRE findings will be independently interpreted by two radiologistsThe role of MRE in distinguishing gut tuberculosis from Crohn's disease will be determined.

DETAILED DESCRIPTION:
The clinical presentation of gut tuberculosis and Crohn's disease is very similar. In areas endemic of tuberculosis infection, differentiating the two diseases remains difficult. Both disease entities can have similar clinical, endoscopic and histological findings. Yet, wrongly diagnosing gut tuberculosis as Crohn's disease can potentially result in disastrous outcomes, especially when anti-tumor necrosis factor therapy, an important therapeutic option for Crohn's disease, can result in fulminant reactivation of tuberculosis.

Magnetic resonance enterography (MRE) is emerging as a effective imaging modality in evaluating the disease status of Crohn's disease. MRE, unlike computed tomography, emits no radiation, and is suitable for repeated serial imaging in younger-age populations. Ulcerations, strictures, transmural enhancement and mesenteric combing of the small bowel can be clearly demonstrated via MRE in Crohn's disease. Yet, the utilization of MRE in diagnosing gut tuberculosis remains largely unexplored. Whether MRE can be used to differentiate gut tuberculosis from Crohn's disease remains unknown.

The investigators plan to consecutively recruit 150 patients presenting to our hospital in Shenzhen, China, for new onset of lower gastrointestinal symptoms and ileocecal mucosal lesions of uncertain diagnosis as evidenced by the presence of inflammation, ulceration, strictures or nodules on colonoscopy.All recruited participants will undergo MRE, to be performed on a 1.5 Tesla scanner (Magnetom Avanto, Siemens Healthcare, Erlangen, Germany). MRE findings will be independently interpreted by two radiologists with special expertise in abdominal MR imaging and blinded to the patients' clinical data. The relationship between radiological patterns and clinical, endoscopic and histological findings will be analyzed. The role of MRE in distinguishing gut tuberculosis from Crohn's disease will be determined.

ELIGIBILITY:
Inclusion Criteria:

* New-onset lower gastrointestinal symptoms of less than 3 months
* Ileocecal mucosal lesions of uncertain diagnosis as evidenced by the presence of inflammation, ulceration, strictures or nodules on colonoscopy.
* No prior tuberculosis treatment
* No prior immunomodulatory or anti-tumor necrosis factor treatment

Exclusion Criteria:

* Stage 4 or 5 chronic kidney disease, i.e. a glomerular filtration rate of <=30 ml/min.
* Contraindications to magnetic resonance imaging, including the installation of metallic devices or implants in-situ (e.g. pacemakers)
* Prior intestinal resection
* Known concomitant chronic small / large bowel disease, including ulcerative colitis, eosinophilic gastroenteritis, NSAID-related enterography etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with new-onset of lower gastrointestinal symptoms and ileocecal mucosal lesions of uncertain diagnosis as evidenced by the presence of inflammation, ulceration, strictures or nodules on colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Small / large bowel transmural enhancement | During procedure
  Via magnetic resonance enterography independently interpreted by two radiologist with expertise

SECONDARY OUTCOMES:
Skip lesions in small / large bowel | During procedure
  Via magnetic resonance enterography independently interpreted by two radiologist with expertise
Vascular engorgement | During procedure
  Via magnetic resonance enterography independently interpreted by two radiologist with expertise
Mesenteric combing | During procedure
  Via magnetic resonance enterography independently interpreted by two radiologist with expertise

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Kay Seto, MD, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No